CLINICAL TRIAL: NCT02058004
Title: Does Cricoid Pressure Reduce the Risk of Aspiration?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other)
Responsible Party: Principal Investigator, John (J Kyle) K. Bohman, M.D., Instructor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-003837
Record Dates: First submitted 2014-01-26; First posted 2014-02-07 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Microaspiration; Acute Respiratory Distress Syndrome (ARDS); Hospital Acquired Pneumonia
Keywords: Microaspiration; ARDS; Hospital acquired pneumonia; Cricoid pressure
MeSH Terms: conditions — Respiratory Distress Syndrome; Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cricoid pressure (Experimental): Patients randomized to receive cricoid pressure during endotracheal intubation.
  Interventions: Procedure: Cricoid pressure
- No cricoid pressure (No Intervention): Patients randomized to receive no cricoid pressure during endotracheal intubation.

INTERVENTIONS:
Procedure: Cricoid pressure — Firm pressure on the cricoid cartilage with the goal of occluding the esophagus during endotracheal intubation.
  Arms: Cricoid pressure

SUMMARY:
In modern anesthesia practice, the application of cricoid pressure during intubation is not infrequently used with the goal of preventing gastric-to-pulmonary aspiration. The evidence to support this practice is very scarce, and there have recently been many reports in the literature questioning the safety of cricoid pressure during intubation. Therefore, the goal of this study will be to randomize those at risk for microaspiration to receive cricoid pressure versus no cricoid pressure during intubation. We will specifically exclude those patients thought to be at the highest risk of aspiration (it is considered standard of care to perform cricoid pressure during intubation of this population). We will include those patients with some risk factors for aspiration (it is not considered standard of care to apply cricoid pressure during intubation of this population).

DETAILED DESCRIPTION:
Gastric-to-pulmonary aspiration during induction of anesthesia remains a significant risk in the modern practice of anesthesia.(1) Macroaspiration (grossly visible aspiration) has been clearly associated with severe pulmonary injury.(1-4) More recently, microaspiration (aspiration without grossly visible gastric material) has also been associated with significant morbidity.(2) Specifically, microaspiration has been associated with acute respiratory distress syndrome (ARDS)(5), ventilator associated pneumonia (VAP)(6) and acute respiratory failure due to bronchoconstriction and ventilation-perfusion mismatching. Pepsin A has been shown to be a very specific biochemical marker for gastric-to-pulmonary aspiration.(7) In our previous studies, we demonstrated the rate of microaspiration in normal elective surgical patients without risk factors for aspiration was 4% as detected by the ELISA assay for pepsin A.(8) This compared with a rate of 12.5% in patients with risk factors for microaspiration including obesity, GERD (gastroesophageal reflux disease) and diabetes. One proposed technique to prevent gastric-to-pulmonary aspiration is cricoid pressure. Recently, there has been growing evidence which calls into question the effectiveness of cricoid pressure. Radiologic studies by Smith et al yield indirect evidence to suggest that cricoid pressure may not reliably occlude the esophagus.(9,10) Currently, cricoid pressure for patients with risk factors for microaspiration (obesity, GERD and diabetes) is used commonly but inconsistently.(11) By using the same sampling and analysis techniques employed in our previous microaspiration studies, the currently proposed study will provide a very sensitive and specific assessment of the effectiveness of cricoid pressure to prevent aspiration during elective induction of anesthesia and intubation. Our proposed study would enroll patients with risk factors for microaspiration who are scheduled to undergo high-risk (for pulmonary complications) elective surgery requiring endotracheal intubation. We will exclude those with risk factors for macroaspiration (including bowel obstruction, non-fasting status and esophageal pathology associated with increased risk for macroaspiration such as achalasia and hiatal hernia), because cricoid pressure remains the standard of care for those at risk for macroaspiration at our institution. Those patients enrolled will be randomized to receive cricoid pressure versus no cricoid pressure. Immediately following elective intubation, a sample of tracheal secretions from each patient will be obtained and the pepsin A concentration determined. The primary outcome will be the rate of microaspiration determined by the presence of pepsin A in the trachea. Secondary outcomes of interest will be rates of postoperative pulmonary complications including acute respiratory distress syndrome (ARDS) and hospital-acquired pneumonia (HAP). The findings of this study will provide the most direct evidence yet regarding the effectiveness of cricoid pressure for the prevention of gastric-to-pulmonary aspiration during induction of anesthesia and endotracheal intubation. Ultimately, the findings of this study will improve patient safety by providing accurate prospective evidence regarding the effectiveness and safety of cricoid pressure in this setting, and will further explore the clinical significance of microaspiration.

ELIGIBILITY:
Inclusion criteria:

* Obesity (BMI>30)
* Diabetes mellitus
* Gastroesophageal reflux disease (GERD)
* schedule cardiac, aortic vascular or non-cardiac thoracic procedure

Exclusion criteria:

* emergent surgery
* risk factors for macroaspiration (non-fasting status, bowel obstruction, achalasia, hiatal hernia, esophageal stricture, esophageal diverticulum), altered level of consciousness, known pregnancy
* preoperative ARDS
* preoperative pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Rate of microaspiration | Within 15 minutes of intubation
  Tracheal secretions will be collected and later analyzed for the presence of pepsin A.

SECONDARY OUTCOMES:
Rate of ARDS | Within 7 days of intubation

OTHER OUTCOMES:
Rate of hospital acquired pneumonia | Within 7 days of intubation

CONTACTS AND LOCATIONS:
Overall Officials: John Bohman, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic - Saint Mary's Campus, Rochester, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota